CLINICAL TRIAL: NCT04726319
Title: Family History App in Personalized Medicine (FHAMe): A Pilot Randomized Controlled Trial
Brief Title: Family History App in Personalized Medicine
Acronym: FHAMe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, June Carroll, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20-0270-E
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cancer, Breast; Cancer, Ovarian; Cancer, Colorectal; Cancer, Prostate; Melanoma; Coronary Artery Disease; Diabetes Mellitus, Type 2
Keywords: Family history; Family medicine; Genetics; Personalized medicine
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Melanoma; Coronary Artery Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Matched-paired randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to usual care, patients will be asked to answer questions about any family history through the use of a questionnaire.
  Interventions: Other: FHAMe Intervention
- Usual Care (No Intervention): Patients receive usual care, which consists of health care providers inquiring about and dealing with family history as they would in usual practice.

INTERVENTIONS:
Other: FHAMe Intervention — Patients will receive an invitation email prior to their scheduled clinical visit which includes information about the study, a link to the YouTube patient presentation, and a link to the consent form and questionnaire. Patients will be invited to fill out the questionnaire prior to their appointment. After patients complete the initial questionnaire, physicians will receive an EMR message on the day of patient's clinic visit alerting them that patient family history information is available and to complete the Family History Action Form. They will be prompted to respond to the message which will open the action form and ask what action the provider intends to take with this family history information. The form will then link to management support tools for use during the patient visit. All participants will attend their clinical visit after which they will receive a post-visit electronic survey regarding their clinical visit and whether family history was reviewed with their provider.
  Arms: Intervention

SUMMARY:
A complete family history (FH) may identify persons at high risk for certain conditions. They can be offered genetic testing and life-saving screening and treatment. In practice, complete FH is rarely collected or entered into the electronic medical record (EMR). The Family History Screening Questionnaire is a survey patients complete to tell whether they are at increased risk of specific cancers, heart disease or diabetes. We will test a new way to record FH that includes an app to improve use of FH by family physicians and patients. The strategy includes education for patients and physicians about the importance of FH; patient completion of the FH questionnaire prior to appointments; and prompts in the EMR. We expect this to help family physicians and patients interpret FH and make the best decisions. We will assess the proportion of patients with new EMR FH information. We will explore if the strategy increases appropriate referrals for screening and genetic consultation for those at increased FH risk. We will also obtain patients' and physicians' feedback on this strategy. This new approach may improve FH information exchange between patients and physicians, encourage shared decision-making and reduce cancer deaths and chronic disease burden.

DETAILED DESCRIPTION:
Family history (FH) is one of the cornerstones of medicine, and provides a glimpse of the genetic make-up of a family. Family physicians (FPs) are in an ideal position to identify those at risk of harboring a genetic mutation requiring further genetics assessment. A challenge in the family medicine clinic is obtaining an adequate FH to triage appropriate patients for further assessment and management. Patients with an identified germline mutation have a variety of therapeutic options including prophylactic surgeries and high risk screening for hereditary cancer syndromes, cardiac devices for inherited cardiac conditions, and intensive statin therapy for those with hypercholesterolemia, all of which can be potentially life-saving.

A systematic review showed that the application of systematic tools which enable information gathering, improves FH accuracy and completeness. Patient-completed FH questionnaires are gaining attention with evidence of reasonable completeness and accuracy. However, challenges have been reported in incorporating these tools including uploading FH results into the EMR and into management strategies.

To address the challenge of obtaining an adequate FH and triaging appropriate patients for further assessment and possibly life-saving interventions, we propose to use a simple FH questionnaire, the "Family History Screening Questionnaire", which will be filled out by patients electronically with the results integrated into the EMR to identify families at risk of inherited diseases.

Overarching Research Objectives:

* To evaluate an innovative strategy to collect family history (FH) and improve personalized primary care. Strategies include: a novel Family History Screening questionnaire (FHSQ) (app), provider alerts, seamless integration into the electronic medical record (EMR), electronic clinical decision support through point-of-care tools, and patient and provider education
* Primary objective: to determine if this innovative strategy will increase the proportion of intervention patients that have updated documentation of family history in the EMR.
* Secondary objective: to describe contextual factors that may influence implementation of this family history strategy into primary care. To explore whether the intervention led to increased discussion about FH and resulted in more personalized screening/management.

This study will determine if increasing awareness of the importance of FH and facilitating collection through a novel FH app with physician alerts, integration into the EMR, electronic decision support and resources, is associated with: increased collection of FH in the EMR, FH discussion by patients and clinicians and personalized, risk appropriate screening/management. Development and implementation of this novel FH app and strategy have the potential to improve FH information exchange between patients and primary care providers, facilitate shared decision-making about personalized screening and management based on FH risk, reduce cancer deaths and chronic disease burden and build the foundation for personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* 30-69 years of age

Exclusion Criteria:

* Pregnancy
* Must be patients of staff physicians (i.e. no resident patients)
* Must have email address registered in the OCEAN system

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with new documentation of family history in EMR | 30 days post visit
  The proportion of patients with new documentation of family history in the EMR within 30 days after the visit, compared to patients in control group practices
Positive family history documentation | 30 days post visit
  The proportion of patients in the intervention arm with positive documented family history in the EMR, compared to patients in control group practices
Proportion of patients in each study arm with new documentation of family history in EMR | 6 months
  The proportion of patients with new documentation of family history in the EMR for each study arm as a whole, over the full 6-month period of the study
Proportion of patients, for each consenting clinician, with new documentation of family history in EMR | 1 year
  The proportion of patients with new documentation of family history in the EMR for each consenting clinician, 6 months prior to the intervention and 6 months after
Family history of breast/ovarian/colorectal/prostate cancer | 30 days post visit
  Proportion of patients with documented family history of cancer in the EMR measured through the number of 1st degree relatives
Changes in risk-appropriate screening based on family history | 30 days post visit
  Through the use of UTOPIAN data which is routinely collected and qualitative interviews with family physicians using semi-structured interview guides, we will explore whether the FH strategy enables risk-appropriate screening based on FH, and referral of patients at high FH risk to genetics

SECONDARY OUTCOMES:
Recruitment rate | 6 months
  Rate of practice and participant recruitment during the intervention period
Participation rate | 6 months
  Proportion of patients completing the questionnaire, and providers attending the webinar, reviewing family history, using clinical tools, and having family history discussions with patients
Usage of family history information | 30 days
  Exploring how family history was obtained and used by patients and physicians through questionnaires and qualitative interviews
Attitudes towards the FHAMe intervention | 30 days
  Exploring patient and team experiences and attitudes to the innovation through questionnaires and qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: June Carroll, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No